CLINICAL TRIAL: NCT01053299
Title: Universal Ultrasound-screening for Developmental Dysplasia of the Hip. 5-12 Years Followup of 4 200 Newborns
Brief Title: Universal Ultrasound-screening for Developmental Dysplasia of the Hip in Newborn
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Vestre VikenHF Kongsberg Sykehus (Other)
Responsible Party: Hans Christian Blom and Guro Elbert (researchcooridinator), VestreVikenHF Kongsberg hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: VestreVikenKS 21517
Record Dates: First submitted 2010-01-20; First posted 2010-01-21 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2010-01

CONDITIONS: Developmental Dysplasia of the Hip (DDH)
Keywords: Developmental dysplasia of the hip (DDH); newborn; universal screening; Universal ultrasound-screening for DDH in newborns; The accuracy of ultrasound-recording of the hip in newborns
MeSH Terms: conditions — Developmental Dysplasia of the Hip | interventions — Prospective Studies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- No treatment (Active Comparator): Every child, without exception, born in the peroid 1.2.1998 - 31.12.2006, still alive, will be called for to take a Xray of their hips aimed at comparing the ultrasound-values taken newborn.
  Interventions: Other: open, prospective cohort-study

INTERVENTIONS:
Other: open, prospective cohort-study — Specific measurements from the X-ray to assess the hip status 5-12 years from the born.

SUMMARY:
All newborn from the period 12.1988 to 31.12.2006 During the two last decades, hip ultrasound has gained acceptance as an accurate screening test for developmental dysplasia of the hip (DDH) and for monitoring the development and treatment of the condition. Debate continues over whether DDH that is detected by ultrasonography is necessarily clinically relevant. The diagnostic accuracy of ultrasound imaging for DDH in the screening population has not been investigated adequately. Studies that investigate the natural course of the disorder, the optimal treatment for DDH, and the best strategy for ultrasound screening are needed. Ultrasound screening at birth for DDH in all newborn infants is standard practice in some European countries but not in the United Kingdom, the United States, or Scandinavia. Evidence is insufficient to support or reject general ultrasound screening of newborns for DDH. (N.F.Woolacott etc 2006, systematic review BMJ) At Vestre Viken HF, Kongsberg, Norway, the investigators implemented universal ultrasound screening in 1998. We will present the long term outcome, including radiographs of the hips after 5-12 years.

DETAILED DESCRIPTION:
All the newborn from the period 1.2.1988 to 31.12.2006 will be called for to take an AP X-ray of the pelvis for assessment of their hips. The data compares to the primary ultrasound-recordings taken newborn.

Radiographs of the pelvis: The x-ray examinations will be performed using low-dose technique. Scrotal lead shield will be used in boys, and the girls will be examined during a menstrual period to exclude pregnancy. The examination will include an erect AP view (feet pointing forward, neutral ab-adduction position of the hips) using a film/focus distance of 1.2 m and centred at 2cm proximal to the pubic bone. To standardise the projection, a rotation index between 0.7 and 1.8 (49;50) will be required. Repeat images will be avoided. A tubing containing a contrast medium will be placed in the x-ray field to give the true horizontal level for measurements of leg length discrepancy. The assessment of the images will be done by a specialist in pediatric radiology in another hospital, and blinded for the primary ultrasound-results. In cases of pathology, the patient will be scheduled for an urgent appointment with a paediatric orthopaedic surgeon.

Image analysis: the following measurements will be performed using a validated digitising program (Pedersen et al, J Pediatric Orthopedic 2004):

1. Markers for DDH:

   CE (centre-edge) angle of Wiberg, Refined CE angle (Ogata) Sharp's angle ADR (the acetabular depth ratio, Murray) FHEI (femoral head extrusion index, Heyman and Herndon) The shape of the lateral acetabulum (subjective assessment)
2. Markers for previous avascular necrosis (AVN)

AP:

Femoral head shape (classified as spherical, mildly flattened or flattened). Caput - trochanter height Projected CCD angle Length and width of the femoral neck (Shape of the physis) Leg length (Trendelenburg) In addition Body Mass Index (BMI) for itch child will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* All newborns form the period 1.21998-31.12.2006

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4200 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Specific measurements of the hip out of an AP Xray of pelvis to assess the diagnostic accuracy of ultrasound imaging for DDH in newborns. | 1.5 - 2 years

SECONDARY OUTCOMES:
Assess the outcome of those treated for DDH from birth based on the primary ultrasound-imaging. | 1,5.2 years

CONTACTS AND LOCATIONS:
Overall Officials: Erlend Skraastad, MD, Study Director — Vestre Viken HF
Locations (1):
- VestreViken HF Kongsberg, Kongsberg, Buskerud, Norway